CLINICAL TRIAL: NCT01438463
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Dose Range Finding Study to Identify the Optimal Dose of PURETHAL® Mites SCIT in Patients With House Dust Mites-induced Persistent Allergic Rhinitis/Rhinoconjunctivitis
Brief Title: PURETHAL® Mites Dose Range Finding Study in Patients With Persistent Allergic Rhinitis/Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM/0037
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: non-seasonal allergy; house dust mite; immunotherapy; dose response
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- PURETHAL Mites, 6,667 AU/ml (Experimental)
  Interventions: Biological: PURETHAL Mites 6,667 AU/ml
- PURETHAL Mites, 20,000 AU/ml (Experimental)
  Interventions: Biological: PURETHAL Mites 20,000 AU/ml
- PURETHAL Mites, 50,000 AU/ml (Experimental)
  Interventions: Biological: PURETHAL Mites 50,000 AU/ml
- PURETHAL Mites, 100,000 AU/ml (Experimental)
  Interventions: Biological: PURETHAL Mites 100,000 AU/ml

INTERVENTIONS:
Biological: Placebo — Increasing volumes of placebo, will be administered by subcutaneous injection (starting with 0.05 ml) at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of placebo, are given at 4-weekly intervals.
  Arms: placebo
Biological: PURETHAL Mites 6,667 AU/ml — Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.
  Arms: PURETHAL Mites, 6,667 AU/ml
Biological: PURETHAL Mites 20,000 AU/ml — Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.
  Arms: PURETHAL Mites, 20,000 AU/ml
Biological: PURETHAL Mites 50,000 AU/ml — Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.
  Arms: PURETHAL Mites, 50,000 AU/ml
Biological: PURETHAL Mites 100,000 AU/ml — Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.
  Arms: PURETHAL Mites, 100,000 AU/ml

SUMMARY:
The objective of the present study is to characterize the dose-response relationship of PURETHAL® Mites with a nasal provocation test in order to support the optimal dose in terms of clinical efficacy and safety.

For this purpose 5 groups of 50 patients, suffering from rhinitis or rhinoconjunctivitis due to House Dust Mite Allergy will be treated during 1 year. Before start, after 6 months of treatment and at the end of the study patients will be subjected to a nasal provocation test.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients (male or female) must be ≥ 18 and ≤ 60 years at screening
* Patients with allergic rhinitis or rhinoconjunctivitis for at least 1 year; allergic symptoms related to HDM, with or without concomitant clinically stable controlled mild to moderate asthma (according to GINA classification)
* Patients with a history of concomitant asthma should have a FEV1 > 70% at inclusion. Patients without a history of asthma should have a FEV1 > 70% or a PEF > 80%.
* Positive SPT to HDM D. pter and/or D. far
* Serum specific IgE-test (ssIgE) level for HDM D. pter or D. far at screening
* Positive nasal provocation test for HDM extract at screening

Exclusion Criteria:

* Current clinically relevant symptoms of seasonal rhinitis/rhinoconjunctivitis caused by other allergen(s) than HDM (with a demonstrated positive SPT for this allergen) at the time of inclusion
* Patients sensitized to animals should not be included if they are symptomatic upon exposure and regularly exposed to animals
* Completed allergen-specific immunotherapy (SCIT or SLIT) with HDM within the last 5 years
* Completed unsuccessful allergen-specific immunotherapy (SCIT or SLIT) within the past 5 years
* Allergen-specific immunotherapy (SCIT or SLIT) with other allergens than HDM during the study period
* Any vaccination one week before start of therapy and during the up-dosing phase
* Any anti-IgE therapy within the last 6 months prior to inclusion and during study
* Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
* Active malignancies or any malignant disease in the past 5 years
* A chronic or acute disease that in the opinion of the investigator might place the patient at an additional risk, including but not limited to the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine disorders, clinically significant renal or hepatic diseases, or haematological disorders
* Moderate to severe nasal obstructive diseases such as polyps, septal deviations etc.
* Clinically significant chronic sinusitis or ocular infection
* Diseases with a contra-indication for the use of adrenaline (e.g. hyperthyroidism, glaucoma)
* Use of systemic corticosteroids within 4 weeks of screening
* Treatment with systemic or local b-blockers
* Participation in a clinical study with a new investigational drug within the last 3 months or a biological within the last 6 months prior to the study or during the study
* Pregnancy, lactation or inadequate contraceptive measures (contraceptive measures considered as adequate include appropriate use of oral contraception, i.m. contraception or a contraceptive device)
* Alcohol, drug, or medication abuse within the past year and during study
* Any abnormal laboratory parameter at screening that in the opinion of the investigator is considered clinically relevant
* Lack of co-operation or compliance
* Severe psychiatric, psychological, or neurological disorders
* Patients who are employees of the department, 1st grade relatives, or partners of the investigator
* Expected changes in HDM exposure during the study (avoidance measures, move, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity to House Dust Mite (HDM) allergen assessed by a Nasal Provocation Test | 12 months

SECONDARY OUTCOMES:
Sensitivity to HDM allergen assessed by a Nasal Provocation Test | 6 months
Average Adjusted daily Symptom Score (AAdSS) | last 2 months of treatment
Peak Nasal Inspiratory Flow (PNIF) | at each visit during 1 year treatment
Specific serum IgE, IgG, and IgG4 immunoglobulin concentrations to house dust mite | 6 and 12 months treatment
Local and systemic reactions after injection as a measure of Safety and Tolerability | 24 hours after each injection during 1 year treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, PhD, MD, Study Chair — University Gent, Belgium
Locations (35):
- Austria (2):
  - Univ.-Klinik für Dermatologie und Venerologie, Innsbruck
  - Universitätsklinik für Hals -, Nasen - und Ohrenheilkunde, Innsbruck
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven campus Sint Rafaël, Leuven
  - CHU de Liège, Liège
- Germany (22):
  - HNO-Praxis Dr. Hippke, Berlin
  - Universitätsklinikum Bonn, Bonn
  - HNO-Praxis, Chemnitz
  - Gemeinschaftspraxis Pneumologie und Allergologie Dr. Hans-Christian Blum, Dortmund
  - HNO-Praxis Dr. U. Thieme, Duisburg
  - Medizinisches Versorgungszentrum, Düren
  - Universitätsklinikum Erlangen, Erlangen
  - HNO Gemeinschaftspraxis, Göttingen
  - Pneumologische Praxis Hannover Nordstadt, Hanover
  - HNO Gemeinschaftspraxis, Heidelberg
  - HNO-Praxis, Jülich
  - POIS Leipzig GbR, Leipzig
  - CRS Clinical Research Services Mannheim GmbH, Mannheim
  - CRS Clinical Research Services Möchengladbach GmbH, Mönchengladbach
  - Gemeinschaftspraxis HNO/Allergologie, München
  - Klinikum der Universität München, München
  - Pneumologie Odeonsplatz, München
  - HNO-Praxis, Pirna
  - Praxisgemeinschaft Reiber & Partner, Schorndorf
  - Universitätsklinikum Stuttgart, Stuttgart
  - Hautarztpraxis, Stuttgart
  - Zentrum für Rhinologie und Allergologie, Wiesbaden
- Netherlands (5):
  - EB FlevoResearch, Almere Stad
  - Allergologie Praktijk Arnhem (APA), Arnhem
  - Albert Schweitzer (Amstelwijck), Dordrecht
  - QPS Onderzoekskliniek Universitair Medisch Centrum Groningen, Groningen
  - St. Elisabethziekenhuis, Tilburg
- Spain (3):
  - Hospital Clinico Barcelona, Barcelona
  - Hospital Universitario Germans Trios i Pujol, Barcelona
  - Hospital Universitari Politecnic La Fe, Valencia